CLINICAL TRIAL: NCT04532632
Title: Taste and Smell Impairment in Critically Ill COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Pinar Ay Sayin (Other)
Responsible Party: Sponsor-Investigator, Pinar Ay Sayin, specialist medical doctor, Sisli Hamidiye Etfal Training and Research Hospital
Organization: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Other Study IDs: 3334-02
Record Dates: First submitted 2020-08-28; First posted 2020-08-31 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Smell Disorder; Taste Disorders; Coronavirus Infection
Keywords: Coronavirus disease-19; anosmia; hyposmia; dysgeusia
MeSH Terms: conditions — Olfaction Disorders; Taste Disorders; Coronavirus Infections; COVID-19; Anosmia; Dysgeusia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluating the smell and taste perceptions of patients hospitalized in the intensive care unit with suspicion of Coronavirus disease-19 diagnosis with a survey study

DETAILED DESCRIPTION:
Patients who were treated in the intensive care unit of Şişli Hamidiye Etfal Training and Research Hospital with the diagnosis of Coronavirus disease-19 will be determined by scanning the hospital registry system. It was planned that patients discharged from the intensive care unit would be called by phone and their complaints about smell and taste disorders were evaluated with a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18-80
* Agree to participate in the study
* Patients treated in the intensive care unit with the diagnosis of Coronavirus disease-19

Exclusion Criteria:

* Pre-existing smell and taste impairment
* The patients have no enough cooperation to answer the questionnaire
* Having additional diseases such as dementia and Alzheimer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-80, who were treated in the intensive care unit with the diagnosis of Coronavirus disease-19 and were discharged
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-09 (Actual)

PRIMARY OUTCOMES:
taste and smell impairment | up to 3 months
  incidence of taste and smell impairment in critically ill subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Sisli Etfal Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hopkins C, Surda P, Whitehead E, Kumar BN. Early recovery following new onset anosmia during the COVID-19 pandemic - an observational cohort study. J Otolaryngol Head Neck Surg. 2020 May 4;49(1):26. doi: 10.1186/s40463-020-00423-8. PMID 32366299
- [Background] Sayin I, Yasar KK, Yazici ZM. Taste and Smell Impairment in COVID-19: An AAO-HNS Anosmia Reporting Tool-Based Comparative Study. Otolaryngol Head Neck Surg. 2020 Sep;163(3):473-479. doi: 10.1177/0194599820931820. Epub 2020 Jun 9. PMID 32513096